CLINICAL TRIAL: NCT00556296
Title: A Phase 3, Randomized, Multi-Center, Double-Blind, Parallel-Group, Placebo-Controlled Study of NRP104 in Children Aged 6-12 Years With Attention Deficit Hyperactivity Disorder
Brief Title: Phase 3 Randomized Double-Blind Placebo-Controlled Study of NRP104 in Children Aged 6-12 With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New River Pharmaceuticals (Industry)
Collaborators: Shire (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRP104.301
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: NRP104
- 2 (Experimental)
  Interventions: Drug: NRP104
- 3 (Experimental)
  Interventions: Drug: NRp104
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NRP104 — NRP104 30mg capsule once daily in a.m.
  Arms: 1
Drug: NRP104 — NRP104 50mg capsule once daily in a.m.
  Arms: 2
Drug: NRp104 — NRP104 70mg capsule once daily in a.m.
  Arms: 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
This study is designed to assess efficacy and safety of NRP-104 administered as a daily dose of 30mg, 50mg or 70mg compared to placebo in the treatment of children aged 6-12 years with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of ADHD combined subtype or the predominantly hyperactive-impulsive subtype based on a psychiatric evaluation that reviews DSM-IV criteria
* functioning at age appropriate levels intellectually
* blood pressure measurements within the 95th percentile for their gender, height and age
* ECG results are within the normal range

Exclusion Criteria:

* comorbid psychiatric diagnosis (such as psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder) or other symptomatic manifestations
* history of seizures (exclusive of febrile seizure), a tic disorder, or a family history of Tourette's disorder
* weighs less than 55 lbs (25 kg)or is significantly overweight or obese
* clinically significant ECG abnormality
* documented allergy or intolerance to amphetamines

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2004-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change score from baseline of the ADHD-RS | 4 weeks

SECONDARY OUTCOMES:
Duration of therapeutic responses using the CPRS ADHD Index | At treatment endpoint, separately for morning, afternoon and evening responses
Clinical global impression of severity(CGI-S) and improvement (CGI-I) | Treatment endpoint
Treatment emergent AEs | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suma Krishnan, Study Director — New River Pharmaceuticals

REFERENCES:
- [Result] Biederman J, Krishnan S, Zhang Y, McGough JJ, Findling RL. Efficacy and tolerability of lisdexamfetamine dimesylate (NRP-104) in children with attention-deficit/hyperactivity disorder: a phase III, multicenter, randomized, double-blind, forced-dose, parallel-group study. Clin Ther. 2007 Mar;29(3):450-63. doi: 10.1016/s0149-2918(07)80083-x. PMID 17577466
- [Result] Faraone SV, Spencer TJ, Kollins SH and Glatt SJ. Moderators of Dose-Response Effects of Lisdexamfetamine Dimesylate Treatment in Children With ADHD. Journal of ADHD and Related Disorders 1(3):16-24, 2010
- [Derived] Jain R, Babcock T, Burtea T, Dirks B, Adeyi B, Scheckner B, Lasser R. Efficacy of lisdexamfetamine dimesylate in children with attention-deficit/hyperactivity disorder previously treated with methylphenidate: a post hoc analysis. Child Adolesc Psychiatry Ment Health. 2011 Nov 4;5(1):35. doi: 10.1186/1753-2000-5-35. PMID 22054243
- [Derived] Waxmonsky JG, Waschbusch DA, Glatt SJ, Faraone SV. Prediction of placebo response in 2 clinical trials of lisdexamfetamine dimesylate for the treatment of ADHD. J Clin Psychiatry. 2011 Oct;72(10):1366-75. doi: 10.4088/JCP.10m05979pur. PMID 21367347
- [Derived] Faraone SV, Spencer TJ, Kollins SH, Glatt SJ. Effects of lisdexamfetamine dimesylate treatment for ADHD on growth. J Am Acad Child Adolesc Psychiatry. 2010 Jan;49(1):24-32. doi: 10.1097/00004583-201001000-00006. PMID 20215923
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html